CLINICAL TRIAL: NCT03683901
Title: The Effect of Electrical Stimulation on Impairment of the Painful Post-Stroke Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, John Chae, MD, VP Research Instititute; Chair, Department of PM&R, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB10-00491
Record Dates: First submitted 2018-09-23; First posted 2018-09-25 (Actual); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Electrical stimulation therapy; TENS; t-NMES; Stroke
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Cohort study; single group but with random serial allocation of treatment type
Masking Description: Participant, Investigator, and Outcomes Assessor were masked to the particular stimulation during each range of motion assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TENS/t-NMES/No stimulation (Experimental): TENS stimulation parameters were of a symmetric waveform, a frequency of 100 Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #7) applied for 10 seconds. t-NMES parameters were a symmetric waveform with 2 second ramp-up and 2 second ramp-down, a frequency of 35Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #3). The t-NMES current intensity was set by adjusting the amplitude to yield the strongest contraction of the underlying muscles without initiating pain. Device and electrodes remained in place but no stimulation was delivered over the 10 second interval. Exposed to each stimulation 3 times for each shoulder ROM.
  Interventions: Device: TENS; Device: t-NMES; Other: No stimulation

INTERVENTIONS:
Device: TENS — Electrical Stimulation
  Other Names: Transcutaneous Electrical Nerve Stimulation
Device: t-NMES — Electrical Stimulation
  Other Names: transcutaneous-Neuromuscular Electrical Stimulation
Other: No stimulation — No stimulation

SUMMARY:
Examination of the effects of short-term use of TENS and t-NMES on passive pain-free ROM of the painful post-stroke shoulder. Treatments are compared with no stimulation.

DETAILED DESCRIPTION:
Single cohort, cross-over study. Subjects undergo passive pain-free ROM of the painful post-stroke shoulder under 3 stimulation conditions. The stimulation was delivered by a trained occupational therapist under three conditions: 10 seconds of TENS, 10 seconds of t-NMES, and 10 seconds of no stimulation. Each subject was exposed to each of the three stimulation conditions three times in a computer-generated random sequence for each outcome measure with a 5-minute wash-out period between each stimulation. This protocol is repeated for each of the two passive movements tested, shoulder abduction and shoulder external rotation.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 months post-stroke
* worst shoulder pain in the last week at least 4 on the 0-10 numerical rating scale,
* adequate cognitive ability to be able to rate their pain in the past week

Exclusion Criteria:

* history of tachyarrhythmia with decreased blood pressure
* uncontrolled seizures (defined as more than one per month)
* an implanted electrical device
* uncompensated hemi-neglect

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12-27 (Actual); Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chae, MD, Principal Investigator — MetroHealth Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chantraine A, Baribeault A, Uebelhart D, Gremion G. Shoulder pain and dysfunction in hemiplegia: effects of functional electrical stimulation. Arch Phys Med Rehabil. 1999 Mar;80(3):328-31. doi: 10.1016/s0003-9993(99)90146-6. PMID 10084443
- [Background] Faghri PD, Rodgers MM, Glaser RM, Bors JG, Ho C, Akuthota P. The effects of functional electrical stimulation on shoulder subluxation, arm function recovery, and shoulder pain in hemiplegic stroke patients. Arch Phys Med Rehabil. 1994 Jan;75(1):73-9. PMID 8291967
- [Background] Leandri M, Parodi CI, Corrieri N, Rigardo S. Comparison of TENS treatments in hemiplegic shoulder pain. Scand J Rehabil Med. 1990;22(2):69-71. PMID 2363027
- [Background] Roosink M, Renzenbrink GJ, Buitenweg JR, van Dongen RT, Geurts AC, Ijzerman MJ. Somatosensory symptoms and signs and conditioned pain modulation in chronic post-stroke shoulder pain. J Pain. 2011 Apr;12(4):476-85. doi: 10.1016/j.jpain.2010.10.009. Epub 2010 Dec 17. PMID 21167792
- [Background] Sluka KA, Deacon M, Stibal A, Strissel S, Terpstra A. Spinal blockade of opioid receptors prevents the analgesia produced by TENS in arthritic rats. J Pharmacol Exp Ther. 1999 May;289(2):840-6. PMID 10215661
- [Background] Soo Hoo J, Paul T, Chae J, Wilson RD. Central hypersensitivity in chronic hemiplegic shoulder pain. Am J Phys Med Rehabil. 2013 Jan;92(1):1-9; quiz 10-3. doi: 10.1097/PHM.0b013e31827df862. PMID 23255268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single group cohort study with random serial allocation of treatment type. All participants underwent each of the three stimulation conditions (TENS, t-NMES, no stimulation) three times in a computer-generated random sequence for each outcome measure with a 5-minute wash-out period between each stimulation.
Groups:
- Hemiplegic Shoulder Pain: Cohort study; single group but with random serial allocation of treatment type (TENS/t-NMES/no stimulation)
Period: Overall Study
Arm/Group | Hemiplegic Shoulder Pain
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants underwent all interventions.
Groups:
- TENS/t-NMES/No Stimulation: Electrical Stimulation-TENS: TENS stimulation parameters were of a symmetric waveform, a frequency of 100 Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #7) applied for 10 seconds.
  Electrical Stimulation-t-NMES: t-NMES parameters were a symmetric waveform with 2 second ramp-up and 2 second ramp-down, a frequency of 35Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #3). The t-NMES current intensity was set by adjusting the amplitude to yield the strongest contraction of the underlying muscles without initiating pain.
  No stimulation: Device and electrodes remained in place but no stimulation was delivered over the 10 second interval.
  Exposed to each stimulation 3 times for each shoulder ROM.
Arm/Group | TENS/t-NMES/No Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Months since stroke [Mean (Standard Deviation); unit: months] | 46.8 (42.1)
Right sided stroke [Count of Participants; unit: Participants] | 6
Worst shoulder pain in the last week (0 min-10 max) [Mean (Standard Deviation); unit: units on a scale] | 7.8 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Passive Range of Motion of Shoulder in Shoulder External Rotation
Description: passive range of motion of shoulder in shoulder external rotation as measured with hand-held goniometer
Time Frame: 10 seconds
Population: Cross-over design. All participants underwent all interventions
Measure: Mean (95% Confidence Interval); unit: degrees
Groups:
- TENS: TENS stimulation parameters were of a symmetric waveform, a frequency of 100 Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #7) applied for 10 seconds. Exposed to this arm 3 times for each shoulder ROM.
  TENS: Electrical Stimulation
- t-NMES: t-NMES parameters were a symmetric waveform with 2 second ramp-up and 2 second ramp-down, a frequency of 35Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #3). The t-NMES current intensity was set by adjusting the amplitude to yield the strongest contraction of the underlying muscles without initiating pain. Exposed to this arm 3 times for each shoulder ROM.
  t-NMES: Electrical Stimulation
- No Stimulation: Device and electrodes remained in place but no stimulation was delivered over the 10 second interval. Exposed to this arm 3 times for each shoulder ROM.
  No stimulation: No stimulation
Arm/Group | TENS | t-NMES | No Stimulation
Number analyzed (Participants) | 10 | 10 | 10
degrees | 66.9 [46.9 to 86.8] | 67.4 [49.4 to 85.4] | 69.1 [49.6 to 88.7]

2. Primary Outcome: Passive Range of Motion of Shoulder in Shoulder Abduction
Description: passive range of motion of shoulder in shoulder abduction as measured with hand-held goniometer
Time Frame: 10 seconds
Population: Cross-over design. All participants underwent all interventions
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | TENS | t-NMES | No Stimulation
Number analyzed (Participants) | 10 | 10 | 10
degrees | 87.8 [70.0 to 105.7] | 87.5 [69.8 to 105.1] | 89.6 [73.9 to 105.4]

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Hemiplegic Shoulder Pain: Electrical Stimulation-TENS: TENS stimulation parameters were of a symmetric waveform, a frequency of 100 Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #7) applied for 10 seconds.
  Electrical Stimulation-t-NMES: t-NMES parameters were a symmetric waveform with 2 second ramp-up and 2 second ramp-down, a frequency of 35Hz, and a pulse duration of 300 microseconds (EMPI 300PVTM program PPR #3). The t-NMES current intensity was set by adjusting the amplitude to yield the strongest contraction of the underlying muscles without initiating pain.
  No stimulation: Device and electrodes remained in place but no stimulation was delivered over the 10 second interval.
  Exposed to each stimulation 3 times for each shoulder ROM.
Arm/Group | Hemiplegic Shoulder Pain
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Electrode placement was determined to provide best possible response for the two movements and stimulation types to maintain blinding; however, may have led to a sub-optimal location for either or both types of stimulation. Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No